CLINICAL TRIAL: NCT06019962
Title: Measurement of Pelvic Tilt 6 Weeks Post-Cesarean Delivery
Brief Title: Pelvic Tilt Following Puerperium
Status: Completed | Type: Observational
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal Abouelyazeed Ali, Lecturer of Physical Therapy for Women's Health, South Valley University
Other Study IDs: Pelvic Tilting
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2023-08

CONDITIONS: Pelvic Obliquity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: 21 postpartum women who delivered by cesarean section
  Interventions: Device: digital pelvic inclinometer
- Group B: 21 females who did not experience pregnancy
  Interventions: Device: digital pelvic inclinometer

INTERVENTIONS:
Device: digital pelvic inclinometer — It is a reliable and valid instrument for measuring pelvic tilt angle

SUMMARY:
The slight anterior pelvic tilt is a physiological posture in healthy males and females, however, excessive anterior pelvic tilt is associated with different lumbopelvic discomfort either during gestation or after childbirth.

DETAILED DESCRIPTION:
As pregnant women move from the 1st to the 3rd trimester, they exhibit a notable increase in the angle of pelvic tilting. This may explain the painful pelvic girdle syndrome during gestation which can last for several weeks postpartum.

When women finish their 6 weeks of puerperium, it may be suspected to return in the pelvic tilting angle to its measurements prior to gestation.

ELIGIBILITY:
Inclusion Criteria:

* Women who underwent cesarean delivery
* Women who were classified as having normal or overweight score on body mass index
* Women in their 6-12 weeks postpartum

Exclusion Criteria:

* Women who underwent vaginal delivery
* Women who were obese on the body mass index
* Women with postpartum duration of less than 6 weeks or more than 12 weeks

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — a study in the field of obstetric physiotherapy
Study Population: 42 subjects participated in this study aged between 18 and 34 years old. They were recruited from South Valley University Hospitals and classified into 2 groups equal in their numbers.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2022-01-29 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
pelvic tilt angle | 6-12 weeks after Cesarean delivery
  angle between the line passing from the posterior and anterior superior iliac spines, and the horizontal plane

SECONDARY OUTCOMES:
pelvic torsion | 6-12 weeks after Cesarean delivery
  the calculated numerical degrees when the angle of pelvic tilt on the right side is substracted from its counterpart on the left side

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, South Valley University, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beatty ME, Zook EG, Russell RC, Kinkead LR. Grain auger injuries: the replacement of the corn picker injury? Plast Reconstr Surg. 1982 Jan;69(1):96-102. PMID 7053516
- [Background] Franklin ME, Conner-Kerr T. An analysis of posture and back pain in the first and third trimesters of pregnancy. J Orthop Sports Phys Ther. 1998 Sep;28(3):133-8. doi: 10.2519/jospt.1998.28.3.133. PMID 9742469
- [Background] Chauhan G, Tadi P. Physiology, Postpartum Changes. 2022 Nov 14. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK555904/ PMID 32310364